CLINICAL TRIAL: NCT03754647
Title: Effect of Vitamin C Upon Selective Serotonin Reuptake Inhibitors-treated Obsessive Compulsive Disorder Patients
Brief Title: Effect of Vitamin C Upon SSRI-treated OCD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr.Taslima Akter, MD, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2018/3110
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: OCD
Keywords: Vitamin C; OCD; MDA; RBC Glutathione
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving SSRIs (No Intervention): This group will be receive SSRIs only
- Patients receiving Vitamin C with SSRIs (Active Comparator): This group will be receive vitamin C (500mg) twice daily with SSRIs for 8 weeks
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — One tablet of Vitamin C (500 mg) twice daily with SSRIs for 8 weeks
  Arms: Patients receiving Vitamin C with SSRIs

SUMMARY:
Title:

Effect of Vitamin C upon Selective Serotonin Reuptake Inhibitors (SSRIs) - treated Obsessive Compulsive Disorder (OCD) patients.

Purpose of the study:

This study aims to examine the effect of vitamin C upon Selective Serotonin Reuptake Inhibitors (SSRIs) - treated Obsessive Compulsive Disorder patients.

Method:

It will be a prospective type of interventional study to to assess the effects of vitamin C along with SSRIs upon OCD patients. The study will be conducted in the Department of Pharmacology and Department of Psychiatry, BSMMU, from September 2017 to February 2019. A total of 90 OCD patients will be selected according to inclusion and exclusion criteria. The patients will be divided randomly into 2 groups: group A and group B. Group A will consist of 45 patients who will receive only SSRIs orally daily and group B would consist of 45 patients who will receive vitamin C, 500 mg BID orally daily along with SSRIs for 8 weeks. To see the effects of Vitamin C, Yale-Brown score of obsessive-compulsive disorders (Y-OCD) would be assessed by Yale-Brown Obsessive Compulsive Scale (Y-BOCS) at baseline (before vitamin C administration) and 8 weeks after intervention. Biochemical parameters of oxidative stress markers such as plasma malondialdehyde (MDA), plasma reduced glutathione (GSH) and plasma vitamin C level would also be performed at baseline (before vitamin C administration) and 8 weeks after intervention.

Ethical consideration:

The study will follow the principles of the Declaration of Helsinki and of the World Medical Assembly. Patients will be informed about the study in easy language and then informed consent will be taken. This study has no potential risk to the patients. Confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
Obsessive compulsive disorder (OCD) is the fourth-most common mental disorder. The World Health Organization (WHO) estimated OCD to be among the top 10 causes of years lived with illness related disability by 2020. Various psychological, social, genetic and biochemical factors are presumed to be involved in the etiology of OCD. Researches so far have indicated that free radical induced injuries are involved in the pathology of OCD. A well-known source of antioxidant is Vitamin C, which is easily available, cheap and more powerful regarding antioxidant effects compared to many other natural sources of vitamin C. Until now little study has been performed to observe the effect of vitamin C administration concurrent to the Selective Serotonin Reuptake Inhibitors (SSRIs) in the treatment of OCD. Therefore the present study has been designed to assess the effects of vitamin C along with SSRIs upon OCD patients. The study would be a prospective type of interventional study to be conducted in the Department of Pharmacology and Department of Psychiatry, BSMMU, from September 2017 to February 2019. A total of 90 OCD patients will be selected according to inclusion and exclusion criteria. The patients will be divided randomly into 2 groups: group A and group B. Group A would consist of 45 patients who will receive only SSRIs orally daily and group B would consist of 45 patients who will receive vitamin C, 500 mg BID orally daily along with SSRIs for 8 weeks. Comparison between the two groups will be performed through biochemical parameters of oxidative stress markers such as serum malondialdehyde (MDA), serum reduced glutathione (GSH) and serum vitamin C levels at baseline (before vitamin C administration) and 8 weeks after intervention by vitamin C. Along with the biochemical parameters, Yale-Brown score of obsessive-compulsive disorders (Y-OCD) would also be assessed by Yale-Brown Obsessive Compulsive Scale (Y-BOCS).Data would be analyzed by Scientific Package for Social Science(SPSS) and represented by tables and figures as applicable. Significance level would be set at 0.05, 0.01 and 0.001. Patient's data will be recorded in a predetermined data sheet. Patients will be informed about the study in easy language and then informed consent will be taken. This study has no potential risk to the patients. Hence, this study would be the first to examine the efficacy of vitamin C as an adjunct to SSRIs in the treatment of OCD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OCD diagnosed by Psychiatry Department of BSMMU.
* OCD patients fulfills Diagnostic criteria of DSM-5.
* Insufficient or depleted plasma Vitamin C level 0.2-0.39 mg/dl or 11-28 µmol/L.
* Patients with YBOCS score more than 14.

Exclusion Criteria:

* Any physical or systemic illness / handicaps.
* Alcohol or substance abuse or dependence.
* Patients with Diabetes, Malignancy, Renal or Hepatic diseases.
* Patients receiving antidepressants within last 2 months.
* Patients with other psychological disorder (such as schizophrenia, bipolar disorder).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-02-10 (Estimated); Study Completion 2019-02-10 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of vitamin C upon Selective Serotonin Reuptake Inhibitors (SSRIs) - treated Obsessive Compulsive Disorder patients. | 8 weeks
  To assess the clinical improvement of OCD patients by Yale-Brown Obsessive Compulsive Scale (Y-BOCS) and compare plasma MDA, RBC glutathione, plasma vitamin C levels at baseline and after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh